CLINICAL TRIAL: NCT01880840
Title: Randomized Trial of the Safety of Astepro 0.15% Nasal Spray and Astepro 0.1% Nasal Spray in Children Ages >6 Months to <6 Years With Allergic Rhinitis
Brief Title: Safety of Astepro 0.15% Nasal Spray and Astepro 0.1% Nasal Spray in Children Ages >6 Months to <6 Years With AR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Collaborators: Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP 442
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2014-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — azelastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astepro 0.15% Nasal Spray (Active Comparator): Nasal Spray at a dosage of 1 spray per nostril twice daily
  Interventions: Drug: 205.5 mcg of azelastine hydrochloride
- Astepro 0.1% Nasal Spray (Active Comparator): Nasal Spray at a dosage of 1 spray per nostril twice daily
  Interventions: Drug: 137 mcg of azelastine hydrochloride

INTERVENTIONS:
Drug: 205.5 mcg of azelastine hydrochloride — nasal spray
  Other Names: astepro .15%
  Arms: Astepro 0.15% Nasal Spray
Drug: 137 mcg of azelastine hydrochloride — nasal spray
  Other Names: astepro .1%
  Arms: Astepro 0.1% Nasal Spray

SUMMARY:
The purpose of this study is to compare the safety of 2 different doses of the investigational use of an allergy medication (Astepro Nasal Spray) in the treatment of allergic rhinitis (AR). This is an open-label study; that is, parent and child will know which group each is in.

DETAILED DESCRIPTION:
Approximately 200 subjects, between the ages of ≥ 6 months to < 6 years of age who have a history of AR will participate in this study.

The study will be conducted at about 20 research centers in the United States. Each research center will enroll approximately 2 to 10 subjects.

The study will involve at least 4 office visits over at least a 4-week period. You will need to keep the appointments as scheduled by the study personnel.

Some medications or therapies could interfere with the safety evaluations conducted in this study. If your child is currently taking any of these medications or therapies, they will need to discontinue them in order to be eligible for this study. Your study doctor will discuss this with you along with information on how this could affect your child's health. If you and the study doctor decide this is appropriate, there is a specific time period that these will need to be discontinued before your child can proceed in study evaluation.

If your child is eligible for study participation, he/she will be randomly assigned (by chance, like the flip of a coin) to one of the following two study drug groups:

* Astepro (azelastine hydrochloride) 0.15% Nasal Spray, 822 mcg (total daily dose); OR
* Astepro (azelastine hydrochloride) 0.1% Nasal Spray, 548 mcg (total daily dose)

The following are being performed for the purposes of this study and are not considered standard care:

* Your child will be placed in one of the two study drug groups by chance.
* You will complete questionnaires about your child's allergy symptoms.
* You will complete diary cards each morning recording your child's allergy symptoms over the previous 24 hours.
* Your child will have his/her vital signs measured (blood pressure, pulse, temperature and breathing rate).
* You and your child will be asked questions regarding your child's use of any medication or supplements and how your child has felt since his/her last visit.
* Blood and urine samples will be collected to assess the safety of taking the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects >6 months to <6 years, inclusive at the screening visit
* A history of AR
* The parent must provide written informed consent and the child must provide assent, if possible
* Willing and able to comply with the study requirements
* May benefit from treatment with Astepro Nasal Spray, based on the Investigator's assessment (based on medical history, physical examination, etc.) of the subject's clinical condition, at both the Screening and Randomization Visits
* General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer
* Subjects receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimen following a brief period of missed injections do not preclude participation)

Exclusion Criteria:

* On nasal examination, subjects with superficial nasal mucosal erosion, moderate nasal mucosal erosion, nasal mucosal ulceration, nasal septum perforation
* Other nasal disease(s) likely to affect deposition of intranasal medication, such as acute sinusitis, rhinitis medicamentosa or clinically significant polyposis or nasal structural abnormalities
* Nasal surgery or sinus surgery within the previous year
* Chronic sinusitis
* The use of any investigational drug within 30 days prior to Visit 1. No investigational products are permitted for use during the conduct of this study
* Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose (Splenda® brand sweetener)
* Respiratory tract infections within two weeks prior to Visit 1.
* Subjects with significant pulmonary disease including asthma. Subjects with intermittent asthma who only require short-acting inhaled bronchodilators are eligible for enrollment. Asthma (with the exception of intermittent asthma). Subjects with intermittent asthma who only require short-acting inhaled bronchodilators (not more often than twice per week) and who do not have nocturnal awakening as a result of asthma are eligible for enrollment
* Chronic obstructive sleep apnea syndrome (clinical diagnosis)
* Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug or that might significantly affect the subject's ability to complete this trial
* Clinically relevant abnormal physical findings or laboratory results which, in the opinion of the investigator, would interfere with the objectives -- Family members of research center or private practice personnel who are directly involved in this study are excluded
* Members of the same family cannot enroll in the study at the same time.
* Subjects who have used medications or therapies that could interfere with safety evaluations (see Section 4.0)
* Any behavioral condition which could affect subject's ability to accurately report symptoms to the caregiver such as developmental delay, attention deficit disorder, and autism

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 191 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Clinical Research Center of Alabama,LLC, Birmingham, Alabama
  - Little Rock Allergy and Asthma Clinical research Center, Little Rock, Alaska
  - West Coast Clinical Trials, Costa Mesa, California
  - Southern California Research, Mission Viejo, California
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - National Allergy, Asthna & Urticaria Centers of Charleston Pa, Charleston, Pennsylvania
  - Texas Allergy Research Center, Dallas, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Paul H Ratner,MD, San Antonio, Texas
  - Live Oak Allergy and Asthma Clinic, San Antonio, Texas
  - Allergy and Asthma Center, Waco, Texas
  - Pediatric Allergy,Asthma and Immunology/Allergy& Asthma care of Waco, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Astepro 0.15%: azelastine hydrochloride 822mcg nasal spray
- Astepro 0.1%: azelastine hydrochloride 548 mcg nasal spray
Period: Overall Study
Arm/Group | Astepro 0.15% | Astepro 0.1%
Started | 95 | 96
Completed | 87 | 91
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Astepro 0.15% Nasal Spray | Astepro 0.1% Nasal Spray | Total
Number analyzed (Participants) | 95 | 96 | 191
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 95 | 96 | 191
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.29 (1.538) | 3.37 (1.595) | 3.33 (1.566)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 45 | 81
  Male | 59 | 51 | 110
Region of Enrollment [Number; unit: participants]
  United States | 95 | 96 | 191

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: The objective of this clinical trial is to evaluate the safety of Astepro 0.15% Nasal Spray and Astepro 0.1% Nasal Spray at a dosage of 1 spray per nostril twice daily in subjects ≥6months to <6 years of age with allergic rhinitis.
  Safety will be assessed on the basis of reported adverse experiences, nasal examinations, laboratory evaluations, and vital signs assessments.
  Data for each age strata will be summarized separately as well as combined.
Time Frame: one month of treatment
Measure: Number; unit: adverse events
Arm/Group | Astepro 0.15% Nasal Spray | Astepro 0.1% Nasal Spray
Number analyzed (Participants) | 95 | 96
adverse events | 43 | 39

ADVERSE EVENTS:
Arm/Group | Astepro 0.15% Nasal Spray | Astepro 0.1% Nasal Spray
Serious Adverse Events (participants affected / at risk) | 1/95 | 0/96
Other Adverse Events (participants affected / at risk) | 23/95 | 15/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astepro 0.15% Nasal Spray (N=95) | Astepro 0.1% Nasal Spray (N=96)
exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — recovered/resolved
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Astepro 0.15% Nasal Spray (N=95) | Astepro 0.1% Nasal Spray (N=96)
pyrexia (General disorders) | 6 | 5
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
sneezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0
dysgusia (Gastrointestinal disorders) | 2 | 0
rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
upper respiratory tract infection (Infections and infestations) | 2 | 1
vomiting (Gastrointestinal disorders) | 2 | 1
otitis media (Ear and labyrinth disorders) | 0 | 3
dermatitis,contact (Skin and subcutaneous tissue disorders) | 0 | 2
oropharyngial pain (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No